CLINICAL TRIAL: NCT00369096
Title: Randomized, Controlled and Open Study to Assess the Efficacy (Peritoneal Biocompatibility) of the Addition of Bemiparin to Icodextrin Solution in Patients in Peritoneal Dialysis With Peritoneal Transport Disorders
Brief Title: Efficacy Study of the Addition of Bemiparin to Icodextrin Solution in Peritoneal Dialysis Patients (Bemidextrina)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Renal Iñigo Alvarez De Toledo (Other)
Collaborators: Infociencia S.L (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRIAT-BEM-2005-01; BEMIDEXTRINA; EudraCT:2005-005695-32
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Peritoneal Diseases
Keywords: Peritoneal Dialysis; Bemiparin; Icodextrin; Peritoneal Transport Disorders
MeSH Terms: conditions — Peritoneal Diseases | interventions — bemiparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bemiparin 3500 IU/day

SUMMARY:
The purpose of this study is to evaluate whether addition of bemiparin, once daily in icodextrin solution for peritoneal dialysis for 16 weeks, increases the peritoneal capacity for ultrafiltration and/or reduces creatinine transport in peritoneal dialysis patients presenting functional disorders related to ultrafiltration deficit and/or high transport.

DETAILED DESCRIPTION:
Peritoneal dysfunction is a common complication in patients in stable treatment with peritoneal dialysis. This peritoneal dysfunction is defined by an elevated creatinine transport and lowered standardized ultrafiltration capacity. The aim of this study is to evaluate the efficacy of the addition of bemiparin to icodextrin solution in patients in peritoneal dialysis with peritoneal transport disorders. The eligible patients are randomly assigned to receive the icodextrin solution with bemiparin or icodextrin solution without bemiparin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old, of either sex, who have given their informed consent to participate in the study.
2. Patients in stable treatment with peritoneal dialysis for more than 6 weeks who present peritoneal dysfunction defined by capacity for standardized ultrafiltration (3.86% glucose maintained in the peritoneum for 4 hours) less than 600 ml and/or elevated creatinine transport (defined by D/P of creatinine higher than 0.65 after 4 hours).
3. Patients treated with icodextrin solution for peritoneal dialysis for at least one month before their inclusion.
4. Patients in whom the remaining dialyzing liquids used in their PD contain glucose and GDP (glucose degradation products).

Exclusion Criteria:

1. Peritonitis in the past 2 months.
2. Patients with bleeding at the time of inclusion, or patients with a history of clinically evident bleeding episodes and/or with increased bleeding due to any other homeostatic alteration that contradicts anticoagulant treatment and/or in the past two months have presented at least one of the following situations: active hemorrhaging or organic lesions susceptible to bleeding (e.g. active peptic ulcer, hemorrhagic cerebrovascular accident, or aneurysms).
3. Major surgery in the past month.
4. Known hypersensitivity to low molecular weight heparin (LMWH), heparin or substances of porcine origin.
5. Known hypersensitivity to icodextrin.
6. Patients treated with systemic anticoagulation.
7. Patients with congenital or acquired bleeding diathesis.
8. Damage to, or surgical interventions of, the central nervous system, eyes or ears within the past 2 months.
9. Acute bacterial endocarditis or slow endocarditis.
10. Patients with a history of heparin-associated thrombocytopenia.
11. Patients with hepatic insufficiency (with values of AST and/or ALT > 5 times the normal value established in the reference range of the local hospital laboratory).
12. Severe arterial hypertension (systolic blood pressure over 200 mmHg and/or diastolic blood pressure over 120 mmHg).
13. Patients with inability or suspected inability to comply with treatment and/or complete the study.
14. Patients who are participating in another clinical trial or have done so in the past 30 days.
15. Patients with a life expectancy less than 6 months.
16. Women who are pregnant, breast-feeding or fertile women who are not using an effective contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: Peritoneal function defined according to the standardized ultrafiltration capacity and/or estimated peritoneal creatinine transport estimated by D/P and mass transfer coefficient during randomized treatment

SECONDARY OUTCOMES:
Safety: Incidence of peritonitis during the randomized treatment period, defined by a cell count of peritoneal effluent with more than 100 leukocytes per mm3 with 50% or more polymorphonuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Selgas Gutierrez, MD, Principal Investigator — Hospital Universitario La Paz; Mª Auxiliadora Bajo Rubio, MD, Principal Investigator — Servicio de Nefrología del Hospital Universitario La Paz (Madrid-Spain); Dra. Gloria del Peso Gilsanz, MD, Principal Investigator — Servicio de Nefrología del Hospital Universitario La Paz (Madrid - Spain); Antonio Carlos Fernández Perpén, MD, Principal Investigator — Servicio de Nefrologia del Hospital Universitario La Princesa (Madrid-Spain); Mercedes L. Velo Plaza, MD, Principal Investigator — Servicio de Nefrologia del Hospital Universitario Príncipe de Asturias de Alcala de Henares (Madrid - Spain); Miguel Pérez Fontán, MD, Principal Investigator — Servicio de Nefrologia del Hospital Juan Canalejo (La Coruña - Spain); Maite Rivera Gorrín, MD, Principal Investigator — Servicio de Nefrologia del Hospital Universitario Ramón y Cajal (Madrid - Spain); MªTeresa Tenorio Cañamas, MD, Principal Investigator — Servicio de Nefrologia del Hospital Universitario Ramón y Cajal (Madrid - Spain); José Portolés Pérez, MD, Principal Investigator — Servicio de Nefrología de la Fundación Hospital de Alcorcón (Madrid - Spain); Juan Manuel López Gómez, MD, Principal Investigator — Servicio de Nefrologia del Hospital Gregorio Marañón (Madrid - Spain); Josep Teixidó, MD, Principal Investigator — Servicio de Nefrologia del Hospital German Trias i Pujol de Badalona (Barcelona-Spain); Mercé Borras, MD, Principal Investigator — Servicio de Nefrologia del Hospital Arnau de Vilanova (Lleida - Spain); Cristina Pérez Melon, MD, Principal Investigator — Servicio de Nefrología del Hospital de Orense(Galicia-Spain); Silvia Ros Ruíz, MD, Principal Investigator — Servicio de Nefrologia del Hospital Regional Universitario Carlos Haya (Málaga-Spain); Teresa González Alvarez, MD, Principal Investigator — Servicio de Nefrología del Hospital de Bellvitge (Barcelona-Spain); Jorge Bartolome, MD, Principal Investigator — Servicio de Nefrologia del Hospital Vall d'Hebron (Barcelona - Spain); Esther Ponz, MD, Principal Investigator — Servicio de Nefrología de la Corporación Sanitaria Parc Taulí (Barcelona - Spain); Pere Torguet, MD, Principal Investigator — Servicio de Nefrologia del Hospital Josep Trueta (Gerona - Spain); Manel Vera i Rivera, MD, Principal Investigator — Servicio de Nefrologia del Hospital Clinic de Barcelona (Barcelona - Spain); Juan Carlos Alonso, MD, Principal Investigator — Servicio de Nefrología del Hospital Lluis Alcanyis Xátiva (Valencia - Spain); Jose Manuel Gil, MD, Principal Investigator — Servicio de Nefrología del Complejo Hospitalario de Jaen (Jaen - Spain)
Locations (17):
- Spain (17):
  - Hospital Regional Universitario Carlos Haya, Málaga, Andalusia
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Corporación Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Hospital Dr. Josep Trueta, Girona, Catalonia
  - Hospital de Orense, Ourense, Galicia
  - Complejo hospitalario de Jaen, Jaén, Jaen
  - Hospital Juan Canajelo, A Coruña
  - Hospital Universitario Príncipe de Asturias, Alcala de Henares (Madrid)
  - Hospital German Trias i Pujol, Badalona (Barcelona)
  - Hospital de Bellvitge, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitario La Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Fundación Hospital Alcorcón, Madrid